CLINICAL TRIAL: NCT06266377
Title: AUT-MENU: Improving Meal Experience of Subjects With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pavia (Other)
Collaborators: Consiglio per la ricerca in agricoltura e l'analisi dell'economia agraria (CREA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11122023
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Food selectivity; Nutrition; Autism spectrum disorder; Collective catering; Food acceptance; mealtime; sustainability
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Non-randomized multi-center intervention with a single arm. Study participants will receive new adapted canteen menus according to the nutritional and sensory needs of the target population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Children afferent to the elementary school where Milano Ristorazione delivers meals and adolescents and young adults enrolled in the State Agricultural Technical Institute Giuseppe Garibaldi (Rome) and Institute I.P.S.E.O.A. "Tor Carbone - A. Narducci."
  Interventions: Other: Administration of menus of collective catering adapted to the sensory and nutritional needs of subjects with Autism Spectrum Disorder; Other: Nutrition education course aimed at caregivers of individuals with Autism Spectrum Disorder

INTERVENTIONS:
Other: Administration of menus of collective catering adapted to the sensory and nutritional needs of subjects with Autism Spectrum Disorder — The AUT-MENU intervention study will be structured in two phases: a preliminary observation phase (T0), which will assess and describe the acceptance of standard meals in the context of collective catering in primary and high schools by the subjects enrolled in the study; and an intervention phase (T1) in which the acceptance of menus targeted to the nutritional and sensory needs of the same subjects enrolled at T0 will be assessed.
  The revision of the standard menus will be carried 1) balancing energy and macronutrient content, 2) promoting adequate weekly food frequencies consumption and portions, to provide an adequate and sustainable menus 3) adapting the sensory characteristics of the foods offered to the sensory needs of individuals with ASD.
  The acceptance of the targeted menus by the enrolled population will be evaluated through meal evaluation forms. These results will be compared with the ones collected during the first observational phase (T0).
Other: Nutrition education course aimed at caregivers of individuals with Autism Spectrum Disorder — A population subgroup will also be selected whose caregivers will be invited to participate in a nutrition education course with the aim of providing parents of subjects with ASD, with knowledge tools to learn how to identify, manage and reduce their children's attitudes of food selectivity.

SUMMARY:
The main goal of this multi-center interventional study is to improve the meal experience of children and adolescents with autism spectrum disorder trough the development of menus for collective catering targeted to their nutritional and sensory needs and the drafting of nutritional indications that can be a reference for collective catering nationwide. After an initial assessment of participants' consumption of meals in the collective service, menus adapted to their nutritional and sensory needs will be administered, and consumption between the initial and adapted menus will be compared. A population subgroup will also be selected whose caregivers will be invited to participate in a nutrition education course with the aim of providing parents of subjects with ASD, with knowledge tools to learn how to identify, manage and reduce their children's attitudes of food selectivity.

DETAILED DESCRIPTION:
The AUT MENU project is a multi-center interventional study conducted on children and adolescents with Autism Spectrum Disorder (ASD) in Milan and Rome.

The main objective of the AUT-MENU project is to improve the meal experience of individuals with Autism Spectrum Disorder (ASD) by developing and disseminating customized menus based on specific dietary recommendations, via collective catering services in schools. The dietary recommendations consider the nutritional and sensory food needs of this population (10.1007/s40519-023-01590-z).

As secondary objective the researchers will evaluate the effect of a nutrition education intervention to the caregivers of the individuals with ASD participating in the study, on reducing their food selectivity. The feasibility of the nutrition education intervention will also be evaluated.

The AUT MENU study deliverable are 1) the development of targeted canteen menus for adults with ASD, according to the nutritional and sensory needs; 2) the elaboration of dietary recommendations to customize canteen menus nutritional and sensory needs for individuals with ASD 3) the development of a nutrition education course aimed at caregivers of a subgroup of the participants.

A total of 16 meal evaluation forms for each participant will be collected on 2 non-consecutive weekly days (for a total of 8 weeks). Both the qualitative and quantitative forms will be filled out by qualified operators, previously trained who assist the participants on a daily basis during lunches eaten at school. For the quantitative evaluation of food consumption, a score will be assigned to the four possible amounts of dish consumed: zero consumption, ¼ of the plate, ½ of the plate, ¾ of the plate, the whole dish.

The nutrition education course aimed at caregivers will be developed in 6 modules. Before and after the course, caregivers will be asked to fill out:

* a questionnaire regarding their children's adherence to the Mediterranean diet
* a validated questionnaire to evaluate their children food selectivity
* a Nutrition Knowledge Questionnaire
* a Satisfaction Questionnaire (of the course)

ELIGIBILITY:
Inclusion Criteria:

* age 5-19 years
* Diagnosis of autism spectrum disorder (grade 1-2 or grade 3)
* Informed consent signed by their caregivers

Exclusion Criteria:

* Subjects who are not autonomous in feeding themselves;
* Presence of neurodevelopmental disorders and/or pathological conditions that require the use of special diets;

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Food acceptance of canteen menus by individuals enrolled in the study | 8 weeks (T0); 8 weeks (T1)
  Meal evaluation forms (score range for each item: 0-1; the score number is directly proportional to the amount of the dish consumed)

SECONDARY OUTCOMES:
Reduction in food selectivity as a result of the targeted nutrition education course | 8 weeks
  Caregivers of a subgroup of the enrolled subjects will undergo a nutrition education course adapted to the needs of individuals with autism spectrum disorder. Caregivers will be asked to fill out questionnaires assessing food selectivity and adherence to the Mediterranean diet before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, MD, Principal Investigator — University of Pavia
Locations (3):
- Italy (3):
  - Milano Ristorazione S.p.A., Milan
  - Istituto I.P.S.E.O.A. "Tor Carbone - A. Narducci"., Roma
  - Istituto Tecnico Agrario Statale "Giuseppe Garibaldi", Roma

REFERENCES:
- [Background] Conti MV, Breda C, Basilico S, Luzzi A, Voto L, Santero S, De Filippo G, Cena H. Dietary recommendations to customize canteen menus according to the nutritional and sensory needs of individuals with autism spectrum disorder. Eat Weight Disord. 2023 Aug 1;28(1):66. doi: 10.1007/s40519-023-01590-z. PMID 37526770
- [Derived] Conti MV, Breda C, Basilico S, Zambon I, Sofroniou A, Ruggeri S, Scalvedi ML, Cena H. Improving Meal Acceptance of Individuals With Autism Spectrum Disorder (AUT-MENU Project): Protocol for a Bicentric Intervention Study. JMIR Res Protoc. 2025 May 21;14:e57507. doi: 10.2196/57507. PMID 40397941